CLINICAL TRIAL: NCT02119585
Title: Observational Study to Analyze Respiratory System Mechanics Changes and Inflammatory Responses During Orthotopic Liver Transplantation (SPPLIT Trial)
Brief Title: Analysis of Respiratory System Mechanics and Inflammatory Response During Orthotopic Liver Transplantation (SPPLIT Trial)
Acronym: SPPLIT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Turin, Italy (Other)
Responsible Party: Principal Investigator, Vito Fanelli MD, PhD, Assistant professor, University of Turin, Italy
Other Study IDs: 0077687
Record Dates: First submitted 2014-04-14; First posted 2014-04-21 (Estimated); Last update posted 2014-12-16 (Estimated); Status verified 2014-12

CONDITIONS: End Stage Liver Diseases
Keywords: orthotopic liver transplantation; ischemia reperfusion syndrome; cytokines; respiratory system elastance; lung elastance; chest wall elastance; shunt; dead space; acute respiratory failure; atelectasis; pleural effusion
MeSH Terms: conditions — Pulmonary Atelectasis; Pleural Effusion

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples at four time points during OLT
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients undergoing OLT: insertion of nasogastric tube for measurements of chest wall mechanics

SUMMARY:
During orthotopic liver transplantation (OLT), respiratory system function may be severely impaired for several reasons including anaesthesia effects, hyperdynamic volume state with fluid overload and ischemia reperfusion injury. In particular, reperfusion syndrome is characterised by the release of several inflammatory mediators such as cytokines and oxygen free radicals which may contribute to alveolar endothelial barrier dysfunction. The object of this study is to investigate the respiratory system mechanics impairment in its partitioning between lung and chest wall.

We hypothesize that impairment of respiratory system mechanics (of both lung and chest wall) occurs after reperfusion phase of liver. This impairment is associated with the systemic inflammatory response following liver reperfusion.

ELIGIBILITY:
Inclusion Criteria:

* orthotopic liver transplantation
* valid informed consent

Exclusion Criteria:

* Age < 18 yrs

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with end stage liver diseases undergoing to liver transplantation
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2014-02; Primary Completion 2014-12 (Estimated); Study Completion 2015-01 (Estimated)

PRIMARY OUTCOMES:
Elastance of Respiratory System, Lung and Chest Wall | at 90 minutes after liver reperfusion
Elastance of Respiratory System, Lung and Chest Wall | at 3 hours after liver reperfusion
Elastance of Respiratory System, Lung and Chest Wall | at 24 hours after liver reperfusion

SECONDARY OUTCOMES:
Acute respiratory failure | 28 days
Ventilator free days | 28 days
ICU length of stay | 28 days
hospital length of stay | 28 days
Inflammatory mediators in plasma samples | baseline, 90 minutes, 3 hours and 24 hours after reperfusion phase
Inflammatory mediators in urine samples | baseline, 90 minutes, 3 hours and 24 hours after reperfusion phase

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda Ospedaliera Città della Salute e della Scienza di Torino, Turin, Turin, Italy